CLINICAL TRIAL: NCT05065372
Title: MANATEE-T1D: Metformin ANd AutomaTEd Insulin Delivery System Effects on Renal Vascular Resistance, Insulin Sensitivity, and Cardiometabolic Function in Youth With Type 1 Diabetes
Acronym: MANATEE-T1D
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kalie Tommerdahl (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Colorado, Denver (Other)
Responsible Party: Sponsor-Investigator, Kalie Tommerdahl, Associate Professor of Pediatric Endocrinology, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-3483; K23HL159292 (NIH)
Record Dates: First submitted 2021-09-13; First posted 2021-10-04 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes; Diabetic Kidney Disease; Cardiovascular Diseases; Endothelial Dysfunction; Insulin Sensitivity
Keywords: Type 1 diabetes; Youth; Insulin sensitivity; Cardiovascular function; Diabetic kidney disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies; Cardiovascular Diseases; Insulin Resistance | interventions — Metformin; p-Aminohippuric Acid; Injections; Iohexol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metformin plus automated insulin delivery system (Active Comparator): Some participants with type 1 diabetes using an automated insulin delivery system will be randomized to receive treatment with metformin and will undergo RPF (Aminohippurate Sodium Injections 20%), GFR (Iohexol Inj 300 MG/ML), and insulin sensitivity (hyperinsulinemic-euglycemic clamp) assessments, in addition to assessments of cardiovascular and endothelial function.
  Interventions: Drug: Metformin Hcl 1000Mg Tab; Drug: Aminohippurate Sodium 20 % Injection; Drug: Iohexol 300 Mg/mL Injectable Solution
- Placebo plus automated insulin delivery system (Placebo Comparator): Some participants with type 1 diabetes using an automated insulin delivery system will be randomized to receive treatment with a placebo pill which is identical in appearance to the metformin pill and will undergo RPF (Aminohippurate Sodium Injections 20%), GFR (Iohexol Inj 300 MG/ML), and insulin sensitivity (hyperinsulinemic-euglycemic clamp) assessments, in addition to assessments of cardiovascular and endothelial function.
  Interventions: Drug: Aminohippurate Sodium 20 % Injection; Drug: Iohexol 300 Mg/mL Injectable Solution; Drug: Placebo
- Multiple daily insulin injections or manual insulin pump plus continuous glucose monitor (Other): Participants with type 1 diabetes using multiple daily injections or an insulin pump in manual mode plus a continuous glucose monitor will not be randomized to receive medication treatment but will undergo RPF (Aminohippurate Sodium Injections 20%), GFR (Iohexol Inj 300 MG/ML), and insulin sensitivity (hyperinsulinemic-euglycemic clamp) assessments, in addition to assessments of cardiovascular and endothelial function.
  Interventions: Drug: Aminohippurate Sodium 20 % Injection; Drug: Iohexol 300 Mg/mL Injectable Solution

INTERVENTIONS:
Drug: Metformin Hcl 1000Mg Tab — Agent used to modify insulin sensitivity
  Other Names: Fortamet; Glucophage; Glumetza; Riomet
  Arms: Metformin plus automated insulin delivery system
Drug: Aminohippurate Sodium 20 % Injection — Diagnostic aid/agent used to measure renal plasma flow and calculate renal vascular resistance
  Other Names: Sodium 4-amino hippurate (PAH) injection 20% (2g/10 mL); Para-aminohippurate; Aminohippuric acid
Drug: Iohexol 300 Mg/mL Injectable Solution — Diagnostic aid/agent used to measure glomerular filtration rate
  Other Names: Omnipaque 300
Drug: Placebo — Identical to Metformin Hcl 1000Mg Tab but without metabolic effects
  Arms: Placebo plus automated insulin delivery system

SUMMARY:
Diabetic kidney disease and cardiovascular disease remain the leading causes of morbidity and mortality in people with type 1 diabetes and are exacerbated with longer duration of diabetes and time outside goal glycemic range. Yet, type 1 diabetes is a complex disease with pathophysiology that extends beyond beta-cell injury and insulin deficiency to include insulin resistance and renal vascular resistance, factors that accelerate cardiovascular disease risk. We have shown that metformin improved peripheral insulin sensitivity and vascular stiffness in youth with type 1 diabetes on multiple daily insulin injections or standard insulin pumps. However, metformin's effect on kidney and endothelial outcomes, and the effects of type 1 diabetes technologies, with or without metformin, on any cardiovascular or kidney outcome, remains unknown. Automated insulin delivery systems combine an insulin pump, continuous glucose monitor, and control algorithm to modulate background insulin delivery and decrease peripheral insulin exposure while improving time in target range and reducing hypoglycemia. We hypothesize that automated insulin delivery systems, particularly when combined with metformin, may modulate renal vascular resistance and insulin sensitivity, thereby impacting cardiometabolic function. MANATEE-T1D is a randomized, double-blind, placebo-controlled trial of 4 months of metformin 2,000 mg daily in 40 youth aged 12-25 years with type 1 diabetes on automated insulin delivery systems vs. 20 control youth with type 1 diabetes on multiple daily injections plus a continuous glucose monitor or an insulin pump in manual mode plus a continuous glucose monitor which will assess for changes in calculated renal vascular resistance and gold standard measures of whole-body and adipose insulin sensitivity, arterial stiffness, and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* T1D and using an automated insulin delivery system or multiple daily insulin injections/manual insulin pump plus continuous glucose monitor for > 6 months
* Age 12-25 years
* Use of an automated insulin delivery system or multiple daily insulin injections plus a continuous glucose monitor or an insulin pump in manual mode plus a continuous glucose monitor for > 6 months
* Hemoglobin A1c < 11%
* No recent episodes of diabetic ketoacidosis (DKA) or hyperglycemic hyperosmolar syndrome (HHS) (within 30 days)
* Pubertal (Tanner stage ≥ 2)
* Weight > 54 kg and BMI > 5th percentile for age and sex

Exclusion Criteria:

* Blood pressure > 140/90 mm Hg
* Hemoglobin < 9 g/dL
* Estimated glomerular filtration rate < 60 mL/min/1.73 m2 or serum creatinine > 1.2 mg/dL or history of urinary albumin to creatinine ratio ≥ 300mg/g or history of acute kidney injury
* Use of anti-diabetic agents except insulin, angiotensin converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARB's), diuretics, daily non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin, sulfonamides, procaine, thiazosulfone or probenecid
* Seafood or iodine allergy
* Pregnancy or breast feeding for females

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Renal vascular resistance | 4 months
  Renal plasma flow will be measured by para-aminohippurate clearance and used to calculate renal vascular resistance
Glomerular filtration rate | 4 months
  Measured by iohexol clearance

SECONDARY OUTCOMES:
Arterial stiffness | 4 months
  Measured by SphygmoCor
Insulin sensitivity | 4 months
  Measured by hyperinsulinemic-euglycemic clamp

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital Colorado/University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided